CLINICAL TRIAL: NCT05274022
Title: Rehabilitation Strategies to Improve Outcomes For Patients With a Lower Extremity Fracture
Acronym: RIFLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brian W. Noehren (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Brian W. Noehren, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 65286; CDMRP-CDMRP-OR200133-A (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2021-11-29; First posted 2022-03-10 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Femoral Fracture; Tibial Fractures
Keywords: Surgical fixation; High intensity interval training
MeSH Terms: conditions — Femoral Fractures; Tibial Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care Physical Therapy Program (Placebo Comparator): Standard of care will follow best practice. The subjects and their physical therapists will be provided with a standardized set of exercises and guidance on what to cover during skilled physical therapy visits.
  Interventions: Other: Standard of Care Physical Therapy Program
- Standard of Care Physical Therapy Program with Speed Walking Intervention (Experimental): Standard of care will follow best practice. The subjects and their physical therapists will be provided with a standardized set of exercises and guidance on what to cover during skilled physical therapy visits. Additionally, subjects will complete the speed walking intervention. Participants will perform at 2 minute warm up followed by 1 minute of walking at their fastest tolerable speed followed by 2 minutes of active recovery where they will walk at a speed of their choosing. The subjects will perform 4 cycles of this followed by a 2 minute cool down at the end.
  Interventions: Other: Standard of Care Physical Therapy Program; Other: Speed Walking Intervention

INTERVENTIONS:
Other: Standard of Care Physical Therapy Program — Standard of care will follow best practice. The subjects and their physical therapists will be provided with a standardized set of exercises and guidance on what to cover during skilled physical therapy visits. As part of the study, all patients will receive the same exercise program. Exercises will include lower extremity strengthening, balance, and mobility exercises with the use of modalities as needed
Other: Speed Walking Intervention — The 4-6 week program will consist of a warm up of active stretching. Following the warm up, subjects will perform a 2 minute warm up followed by 1 minute of walking at their fastest comfortable speed followed by 2 minutes of active recovery where they will walk at a speed of their choosing for 4cycles and then a 2 minute cool down. The program will be performed 12 visits over 4-6 weeks.
  Arms: Standard of Care Physical Therapy Program with Speed Walking Intervention

SUMMARY:
The purpose of this study is to evaluate speed high intensity interval training (HIIT) walking program following an orthopedic trauma.

DETAILED DESCRIPTION:
In HIIT an individual gives short bursts of high effort followed by a longer recovery period.

Increasingly, HIIT style training programs have been used in other clinical populations (heart conditions, kidney failure, severely obese) to yield improved health outcomes and have been shown to be safe and effective. However, this work has not been extended to the orthopedic trauma population. Initiating a treadmill HIIT program during recovery from a lower extremity fracture may prove pivotal to restoring functional abilities, improving strength, and optimizing patient outcomes.

As a starting point to investigate the speed HIIT walking program following an orthopedic trauma, the investigators will focus on femoral and tibial shaft fractures requiring surgical fixation. Subjects will be recruited at a follow-up visit and therefore will not have impaired consent capacity issues at that juncture based on their fracture-related injuries. Even though early postoperative weight bearing has been shown to be safe, there continues to be considerable divergence in recovery after these fractures. For instance, return to work rates for individuals with physical jobs has been reported to be as low as 14% within the first year, resulting in significant stress and financial challenges for the individual. Clearly, improved post-operative rehabilitation strategies are needed for this population.

Aim 1: Assess the feasibility and adherence of the speed HIIT walk program within subjects with a lower extremity fracture.

Primary Hypothesis: 70% of subjects approached about the study will consent and that 80% of subjects will complete the study.

Secondary hypothesis: 80% of subjects will complete all of the treatment sessions and find the treatment (both intervention and standard of care physical therapy) acceptable.

Aim 2: Determine the preliminary effects of the speed HIIT program as compared to the standard of care on patient reported outcomes, functional outcomes and return to work rates, in a pilot randomized control trial.

Primary Hypotheses: Participants in the speed HIIT intervention group will have a significantly higher PROMIS physical function scale as compared to standard of care group at a 6 month follow up.

Secondary hypotheses: Participants in the Speed HIIT intervention group will have higher return to work rates, usual and fastest gait speed, timed step-down test, and 6-minute walk test than the standard of care group at a 6 month follow up.

Tertiary hypothesis: The participants in the speed HIIT program will maintain higher physical function and return to work rates at a 12 month follow up as compared to the standard of care group

Aim 3: Quantify the differences in ground reaction forces, function, psychosocial responses, and patient reported outcomes that occur at the completion of the speed HIIT walk program as compared to the group receiving standard of care physical therapy.

Primary Hypotheses: Participants in the speed HIIT program will be significantly more symmetric in their peak ground reaction force metrics (impulse, loading rates, time, peak values), and have greater self reported physical function, functional outcomes and patient reported outcomes as compared to the standard of care group at the completion of the intervention (19 weeks post hospital discharge).

Secondary hypotheses: Participants completing the speed HIIT program will have greater pain self-efficacy and less fear of movement as compared to the standard of care at the completion of the intervention (19 weeks post hospital discharge) that is maintained at a 6 and 12 month follow up.

Tertiary hypothesis: The participants in the speed HIIT program will maintain higher symmetry in their peak ground reaction force metrics (impulse, loading rates, time, peak values) as compared to the standard of care group at a 6 month follow up.

ELIGIBILITY:
Inclusion Criteria:

* Ability to read and speak English
* Acute orthopedic injury to the femoral or tibial shaft requiring surgical fixation with an intramedullary rod
* Age 18-50 years of age

Exclusion Criteria:

* History of chronic pain defined as pain lasting more than 3 months and bothersome at least half the days over the past 6 months that started before the fracture
* Moderate or severe traumatic brain injury
* Initial treatment requiring amputation
* Not employed at the time of the accident at least 20 hours per week.
* Spinal cord injury
* History of schizophrenia, dementia or neurologic disorder with peripheral dysfunction
* Non ambulatory or limited ability to walk without an assistive device prior to the fracture
* Multiple trauma that prevents early weight bearing
* Current Pregnancy
* Unable to participate in or complete in-person follow-up visits or therapy sessions
* In outpatient Physical Therapy at the start of the intervention
* Use of an assistive device to walk for community ambulation at the 10-12 weeks post hospital discharge time point

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2025-12-18 (Actual); Study Completion 2025-12-18 (Actual)

PRIMARY OUTCOMES:
Self-reported physical function | Up to 12 weeks
  Patient Reported Outcomes Measurement Information System (PROMIS) Physical Function Questionnaire is a 53 question survey with a five point Likert scale ranging from 1 to 5 where a higher number indicates less physical function.
Self-reported physical function | Up to 19 weeks
  Patient Reported Outcomes Measurement Information System (PROMIS) Physical Function Questionnaire is a 53 question survey with a five point Likert scale ranging from 1 to 5 where a higher number indicates less physical function.
Self-reported physical function | 6 months
  Patient Reported Outcomes Measurement Information System (PROMIS) Physical Function Questionnaire is a 53 question survey with a five point Likert scale ranging from 1 to 5 where a higher number indicates less physical function.
Self-reported physical function | 12 months
  Patient Reported Outcomes Measurement Information System (PROMIS) Physical Function Questionnaire is a 53 question survey with a five point Likert scale ranging from 1 to 5 where a higher number indicates less physical function.

SECONDARY OUTCOMES:
60-second step down test | Up to 12 weeks
  Standing on an 4-inch box, participants will step down until the heel gently touches a scale placed on the ground and then return to full knee extension. As many repetitions as possible in 60 seconds will be recorded. Repetitions with over 10% of the body weight registered on the scale will not be counted toward the total number of repetitions completed. The test has previously been shown to have a high interrater reliability of 0.94 and was associated with a change in knee mechanics following an orthopedic surgery.
  Interpretation: More successful repetitions indicate greater neuromuscular control and muscle strength in the lower extremity.
60-second step down test | Up to 19 weeks
  Standing on an 4-inch box, participants will step down until the heel gently touches a scale placed on the ground and then return to full knee extension. As many repetitions as possible in 60 seconds will be recorded. Repetitions with over 10% of the body weight registered on the scale will not be counted toward the total number of repetitions completed. The test has previously been shown to have a high interrater reliability of 0.94 and was associated with a change in knee mechanics following an orthopedic surgery.
  Interpretation: More successful repetitions indicate greater neuromuscular control and muscle strength in the lower extremity.
60-second step down test | 6 months.
  Standing on an 4-inch box, participants will step down until the heel gently touches a scale placed on the ground and then return to full knee extension. As many repetitions as possible in 60 seconds will be recorded. Repetitions with over 10% of the body weight registered on the scale will not be counted toward the total number of repetitions completed. The test has previously been shown to have a high interrater reliability of 0.94 and was associated with a change in knee mechanics following an orthopedic surgery.
  Interpretation: More successful repetitions indicate greater neuromuscular control and muscle strength in the lower extremity.
Usual Gait Speed | Up to 12 weeks
  Participant usual gait speed as measured over 2 trials of walking along a 20 meter walkway at their usual walking speed.
Usual Gait Speed | Up to 19 weeks
  Participant usual gait speed as measured over 2 trials of walking along a 20 meter walkway at their usual walking speed.
Usual Gait Speed | 6 months
  Participant usual gait speed as measured over 2 trials of walking along a 20 meter walkway at their usual walking speed.
Fastest Walking Speed | Up to 12 weeks
  Participant usual gait speed as measured over 2 trials of walking along a 20 meter walkway at their fastest walking speed.
Fastest Walking Speed | Up to 19 weeks
  Participant usual gait speed as measured over 2 trials of walking along a 20 meter walkway at their fastest walking speed.
Fastest Walking Speed | 6 months
  Participant usual gait speed as measured over 2 trials of walking along a 20 meter walkway at their fastest walking speed.
Six-minute walk Test: | Up to 12 weeks
  The participant will be provided with six minutes to walk as far as possible.
Six-minute walk Test: | Up to 19 weeks
  The participant will be provided with six minutes to walk as far as possible.
Six-minute walk Test: | 6 months
  The participant will be provided with six minutes to walk as far as possible.
Pain Assessment | Up to 12 weeks
  Brief Pain Inventory (BPI) will be used to measure pain intensity. This is a four-item scale that measures current, worst, least, and average pain. Each of these four items are measured on a numeric scale from 0 to 10 with 0 being ''no pain'' and 10 being ''severe pain.''
Pain Assessment | Up to 19 weeks
  Brief Pain Inventory (BPI) will be used to measure pain intensity. This is a four-item scale that measures current, worst, least, and average pain. Each of these four items are measured on a numeric scale from 0 to 10 with 0 being ''no pain'' and 10 being ''severe pain.''
Pain Assessment | 6 months
  Brief Pain Inventory (BPI) will be used to measure pain intensity. This is a four-item scale that measures current, worst, least, and average pain. Each of these four items are measured on a numeric scale from 0 to 10 with 0 being ''no pain'' and 10 being ''severe pain.''
Pain Assessment | 12 months
  Brief Pain Inventory (BPI) will be used to measure pain intensity. This is a four-item scale that measures current, worst, least, and average pain. Each of these four items are measured on a numeric scale from 0 to 10 with 0 being ''no pain'' and 10 being ''severe pain.''
Pain self-efficacy scale (PSEQ) | Up to 12 weeks
  The Pain Self-Efficacy Questionnaire (PSEQ) is a 10-item questions and will be used measure an individual's beliefs about their ability to participate in social activity and accomplish their goals despite the presence of pain. PSEQ has demonstrated excellent internal consistency, test-retest reliability, and construct validity.
  Interpretation: Greater self-efficacy (higher survey score) is related to reductions in disability, pain intensity, fear of movement and pain, and affective distress in patients with chronic pain.
  Scale: 0-6 0 (not at all confident)
  1 2 3 4 5 6 (completely confident)
Pain self-efficacy scale (PSEQ) | Up to 19 weeks
  The Pain Self-Efficacy Questionnaire (PSEQ) is a 10-item questions and will be used measure an individual's beliefs about their ability to participate in social activity and accomplish their goals despite the presence of pain. PSEQ has demonstrated excellent internal consistency, test-retest reliability, and construct validity.
  Interpretation: Greater self-efficacy (higher survey score) is related to reductions in disability, pain intensity, fear of movement and pain, and affective distress in patients with chronic pain.
  Scale: 0-6 0 (not at all confident)
  1 2 3 4 5 6 (completely confident)
Pain self-efficacy scale (PSEQ) | 6 months
  The Pain Self-Efficacy Questionnaire (PSEQ) is a 10-item questions and will be used measure an individual's beliefs about their ability to participate in social activity and accomplish their goals despite the presence of pain. PSEQ has demonstrated excellent internal consistency, test-retest reliability, and construct validity.
  Interpretation: Greater self-efficacy (higher survey score) is related to reductions in disability, pain intensity, fear of movement and pain, and affective distress in patients with chronic pain.
  Scale: 0-6 0 (not at all confident)
  1 2 3 4 5 6 (completely confident)
Pain self-efficacy scale (PSEQ) | 12 months
  The Pain Self-Efficacy Questionnaire (PSEQ) is a 10-item questions and will be used measure an individual's beliefs about their ability to participate in social activity and accomplish their goals despite the presence of pain. PSEQ has demonstrated excellent internal consistency, test-retest reliability, and construct validity.
  Interpretation: Greater self-efficacy (higher survey score) is related to reductions in disability, pain intensity, fear of movement and pain, and affective distress in patients with chronic pain.
  Scale: 0-6 0 (not at all confident)
  1 2 3 4 5 6 (completely confident)
Tampa scale of kinesiophobia (TSK) | Up to 12 weeks
  The TSK is a 17-item questionnaire and will be administered to record fear of movement (kinesiophobia).
  Interpretation: Higher survey scores indicates greater kinesiophobia in people with chronic pain.
  Scale: (0-3) 0, Strongly disagree
  1. Disagree
  2. Agree
  3. Strongly agree
Tampa scale of kinesiophobia (TSK) | Up to 19 weeks
  The TSK is a 17-item questionnaire and will be administered to record fear of movement (kinesiophobia).
  Interpretation: Higher survey scores indicates greater kinesiophobia in people with chronic pain.
  Scale: (0-3) 0, Strongly disagree
  1. Disagree
  2. Agree
  3. Strongly agree
Tampa scale of kinesiophobia (TSK) | 6 months
  The TSK is a 17-item questionnaire and will be administered to record fear of movement (kinesiophobia).
  Interpretation: Higher survey scores indicates greater kinesiophobia in people with chronic pain.
  Scale: (0-3) 0, Strongly disagree
  1. Disagree
  2. Agree
  3. Strongly agree
Tampa scale of kinesiophobia (TSK) | 12 months
  The TSK is a 17-item questionnaire and will be administered to record fear of movement (kinesiophobia).
  Interpretation: Higher survey scores indicates greater kinesiophobia in people with chronic pain.
  Scale: (0-3) 0, Strongly disagree
  1. Disagree
  2. Agree
  3. Strongly agree
Return to Work Status: Hours Worked | Up to 12 weeks
  Work Productivity and Activity Impairment Questionnaire (WPAI) part 1 includes three questions about the number of hours worked in the last seven days.
Return to Work Status: Hours Worked | Up to 19 weeks
  Work Productivity and Activity Impairment Questionnaire (WPAI) part 1 includes three questions about the number of hours worked in the last seven days.
Return to Work Status: Hours Worked | 6 months
  Work Productivity and Activity Impairment Questionnaire (WPAI) part 1 includes three questions about the number of hours worked in the last seven days.
Return to Work Status: Hours Worked | 12 months
  Work Productivity and Activity Impairment Questionnaire (WPAI) part 1 includes three questions about the number of hours worked in the last seven days.
Return to Work Status: Ability to Work | Up to 12 weeks
  Work Productivity and Activity Impairment Questionnaire (WPAI) part 2 includes 2 questions with a 10 point scale where a lower number indicates a greater ability to work with no health problems.
Return to Work Status: Ability to Work | Up to 19 weeks
  Work Productivity and Activity Impairment Questionnaire (WPAI) part 2 includes 2 questions with a 10 point scale where a lower number indicates a greater ability to work with no health problems.
Return to Work Status: Ability to Work | 6 months
  Work Productivity and Activity Impairment Questionnaire (WPAI) part 2 includes 2 questions with a 10 point scale where a lower number indicates a greater ability to work with no health problems.
Return to Work Status: Ability to Work | 12 months
  Work Productivity and Activity Impairment Questionnaire (WPAI) part 2 includes 2 questions with a 10 point scale where a lower number indicates a greater ability to work with no health problems.

OTHER OUTCOMES:
Loading of the lower extremity | Up to 12 weeks
  The ground reaction forces of the injured and non injured limb will be evaluated over the course of recovery to assess when loading between limbs becomes symmetric.
Loading of the lower extremity | Up to 19 weeks
  The ground reaction forces of the injured and non injured limb will be evaluated over the course of recovery to assess when loading between limbs becomes symmetric.
Loading of the lower extremity | 6 months
  The ground reaction forces of the injured and non injured limb will be evaluated over the course of recovery to assess when loading between limbs becomes symmetric.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Noehren, Ph.D., Principal Investigator — University of Kentucky
Locations (2):
- United States (2):
  - University of Kentucky, Lexington, Kentucky
  - Vanderbilt University, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-09-16): https://cdn.clinicaltrials.gov/large-docs/22/NCT05274022/ICF_000.pdf